

#### TRIAL STATISTICAL ANALYSIS PLAN

c36670861-01

**BI Trial No.:** 1450-0001

Title: Safety, tolerability, pharmacokinetics, and pharmacodynamics of

single rising intravenous doses of BI 765080 in healthy male subjects (single-blind, randomised, placebo-controlled, parallel-

group design)

Including Protocol Amendment 2 [c31414158-03]

Investigational

**Product:** 

BI 765080

Responsible trial statistician:

Phone: Fax:

Date of statistical

21-Sep-2021 SIGNED

analysis plan:

Version: Final


#### Proprietary confidential information

© 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

| 1. | TABLE OF CONTENTS | |
|---|---|---|
| TITLE 1 | PAGE | 1 |
| 1. | TABLE OF CONTENTS. | 2 |
| LIST O | F TABLES | |
| 2. | LIST OF ABBREVIATIONS | |
| 3. | INTRODUCTION | |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY | 8 |
| 5. | ENDPOINTS | |
| 5.1<br>5.2 | PRIMARY ENDPOINT | |
| 5.2<br>5.2.1 | Key secondary endpoints | |
| 5.2.2 | Secondary endpoints | |
| 01212 | Secondary chaponits | |
| 5.3.1 | Safety parameters | 9 |
| 6. | GENERAL ANALYSIS DEFINITIONS12 | 2 |
| 6.1 | TREATMENTS12 | |
| 6.2 | IMPORTANT PROTOCOL DEVIATIONS | |
| 6.3 | SUBJECT SETS ANALYSED1 | 3 |
| 6.5 | POOLING OF CENTRES | 5 |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS | |
| <b>6.7</b> | BASELINE, TIME WINDOWS AND CALCULATED VISITS1 | |
| 7. | PLANNED ANALYSIS1 | 7 |
| <b>7.1</b> | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS1 | |
| <b>7.2</b> | CONCOMITANT DISEASES AND MEDICATION18 | |
| <b>7.3</b> | TREATMENT COMPLIANCE1 | |
| 7.4 | PRIMARY ENDPOINTS1 | 8 |
| 7.4.1 | | |
| <b>—</b> — | Primary analysis of the primary endpoints1 | 8 |
| 7.5<br>7.5.1 | Primary analysis of the primary endpoints | 8 |
| 7.5.1 | Primary analysis of the primary endpoints | 8<br>8<br>8 |
| 7.5.1<br>7.5.2 | Primary analysis of the primary endpoints | 8<br>8<br>8<br>9 |
| 7.5.1 | Primary analysis of the primary endpoints | 8<br>8<br>8<br>9 |
| 7.5.1<br>7.5.2 | Primary analysis of the primary endpoints | 8<br>8<br>8<br>9 |

TSAP for BI Trial No: 1450-0001 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| 7.7 | EXTENT OF EXPOSURE | 21 |
|--------------|--------------------------------------------|----------|
| <b>7.8</b> | SAFETY ANALYSIS | 21 |
| <b>7.8.1</b> | Adverse Events | 21 |
| 7.8.2 | Laboratory data | 22 |
| 7.8.3 | Vital signs | |
| 7.8.4 | ECG | |
| 7.8.5 | Others | |
| 7.8.5.1 | Physical examination | 25 |
| 7.8.5.2 | Oral body temperature | |
| 7.8.5.3 | Local tolerability assessment | |
| 7.8.5.4 | Body weight | |
| o TIME | | |
| 8. HIVIE | EPOINT OF RELEASE OF TREATMENT INFORMATION | <u> </u> |
| 11. | HISTORY TABLE. | 33 |

# Boehringer Ingelheim TSAP for BI Trial No: 1450-0001 Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# **LIST OF TABLES**

| Table 6.1: 1 | Analysis phases for statistical analysis of AEs, and actual treatment for | |
|---|---|---|
| | analysis of laboratory data, vital signs, ECG and local tolerability | 12 |
| Table 6.3: 1 | Subject sets analyzed | 14 |
| Table 6.7: 1 | Time schedule of 12-lead ECG recordings with centralised evaluation | 16 |
| Table 11: 1 | History table | 33 |

TSAP for BI Trial No: 1450-0001 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### LIST OF ABBREVIATIONS 2.

| Term | Definition / description |
|---|---|
| AE | Adverse Event |
| AESI | Adverse event of special interest |
| ALT | Alanine aminotransferase |
| AST | Aspartate aminotransferase |
| $AUC_{0-\infty}$ | Area under the concentration-time curve of the analyte in serum over the time interval from 0 extrapolated to infinity |
| BI | Boehringer Ingelheim |
| $C_{\text{max}}$ | Maximum measured concentration of the analyte in serum |
| COVID | Coronavirus disease |
| CTP | Clinical Trial Protocol |
| CTR | Clinical Trial Report |
| CV | Arithmetic coefficient of variation |
| ECG | Electrocardiogram |
| ECGPCS | ECG PK concentration set |
| gCV | geometric coefficient of variation |
| gMean | Geometric mean |
| HR | Heart rate |
| ICH | International Conference On Harmonisation |
| IPD | Important protocol deviations |
| LLOQ | Lower limit of quantification |
| MedDRA | Medical Dictionary For Regulatory Activities |
| PD | Pharmacodynamics |
| PK | Pharmacokinetics |
| PKS | Pharmacokinetic parameter analysis set |
| PR | Pulse rate |
| QRS complex | Combination of the Q, R, and S waves |
| QT interval | Time between start of the Q-wave and the end of the T-wave in an electrocardiogram |
| QTcB | QT interval, heart rate corrected according to Bazetts formula |

Boehringer Ingelheim
TSAP for BI Trial No: 1450-0001
Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Term | Definition / description |
|---|---|
| QTcF | QT interval, heart rate corrected according to Fridericias formula |
| RAGe | Report appendix generator |
| RPM | Report Planning Meeting |
| RR interval | ECG interval from the peak of the R wave to the peak of the subsequent R wave |
| SAE | Serious adverse event |
| SD | Standard Deviation |
| SOC | System Organ Class |
| TS | Treated set |
| TSAP | Trial Statistical Analysis Plan |
| ULN | Upper limit of normal range |

## 3. INTRODUCTION

As per ICH E9 (1) the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the revised CTP, and to include detailed procedures for executing the statistical analysis of the primary variables and other data.

This TSAP assumes familiarity with the CTP and its amendments. In particular, the TSAP is based on the planned analysis specification as written in CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the revised CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomisation.

Study data as collected in the eCRF will be stored in a trial database within the RAVE EDC system. All study data also including external data will then be uploaded to the CDR data warehouse.

PK parameters will be calculated using Phoenix WinNonlin<sup>TM</sup> software (version Phoenix 6.3,

TSAP for BI Trial No: 1450-0001 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 4. CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

All analyses described in this TSAP are in accordance with the statistical methods described in the revised CTP.

#### 5. ENDPOINTS

#### 5.1 PRIMARY ENDPOINT

Primary endpoint is the percentage of subjects with drug-related adverse events.

#### 5.2 SECONDARY ENDPOINTS

#### 5.2.1 Key secondary endpoints

Not applicable.

#### 5.2.2 Secondary endpoints

Secondary endpoints are PK endpoints of BI 765080, as defined in Section 2.1.3 of the CTP:

- $AUC_{0-\infty}$  (area under the concentration-time curve of the analyte in serum over the time interval from 0 extrapolated to infinity)
- $C_{max}$  (maximum measured concentration of the analyte in serum)

#### 5.3.1 Safety parameters

Safety and tolerability of BI 765080 will be assessed based on further safety parameters defined in Section 2.2.2.1 of the **CTP**:

- AEs (including clinically relevant findings from the physical examination)
- Safety laboratory tests
- 12-lead ECG
- Continuous ECG monitoring
- Vital signs (blood pressure and pulse rate), oral body temperature
- Local tolerability assessment

#### **Local tolerability**

Local tolerability will be assessed as absence or presence of "swelling", "induration", "heat", "redness", "pain", or "other findings".

#### 12-lead ECG endpoints

For the definition of baseline and a summary of time points please refer to Section 6.7.

#### Quantitative ECG endpoints:

The following quantitative ECG endpoints will be determined for the ECG variables QTcF, QT, HR, PR, QRS, RR and QTcB derived as described in <u>Additional Section 10.1</u>:

- absolute values (per time point)
- changes from baseline (per time point)
- percent changes from baseline (per time point; for HR, PR, QRS)

#### Categorical ECG endpoints

The following categorical ECG endpoints will be determined based on the quantitative ECG endpoints, except for QTcB. QTcB will only be listed.

- New onset (meaning that this or a higher category was not present at baseline) of maximum QTcF interval > 450 to 480 msec, > 480 to 500 msec, or > 500 msec on treatment. For assignment of a particular subject to one of the above categories, all time points on-treatment (refer to Table 6.7: 1) will be considered.
- Maximum change from baseline in QT interval of  $\leq$  60 msec, or > 60 msec on treatment
- Maximum change from baseline in QTcF interval of  $\leq$  30 msec, > 30 to  $\leq$  60 msec, or > 60 msec on treatment

The occurrence of any of the following will be viewed as "notable findings":

- New onset (not present at baseline) of uncorrected QT interval > 500 msec at any time on treatment
- New onset of QTcF interval > 500 msec at any time on treatment
- Change from baseline of QTcF > 60 msec at any time on treatment
- Percent change from baseline of HR  $\geq$  25%, when corresponding on-treatment value of HR is > 100 beats/min, or percent change from baseline of HR  $\leq$  25%, when corresponding on-treatment value of HR is < 50 beats/min, at any time on treatment
- Percent change from baseline of PR  $\geq$  25%, when corresponding on-treatment value of PR interval is > 200 msec, at any time on treatment
- Percent change from baseline of QRS  $\geq$  10%, when corresponding on-treatment value of QRS duration is > 110 msec, at any time on treatment

For a detailed description of 'new onset', refer to Additional Section 10.3.





#### 6. GENERAL ANALYSIS DEFINITIONS

#### 6.1 TREATMENTS

For basic study information on treatments to be administered, assignment of treatment groups, and selection of doses, cf. Section 4 of the CTP.

Subjects will receive a 30 minutes intravenous infusion containing

- powder for solution of either a single dose of 1, 10, 25, 50, 100 or 200 mg of BI 765080 (test treatments)
- a matching placebo (reference treatment)

All placebo subjects will be analysed in one pooled placebo group (i.e. no distinction between dose groups will be made for placebo subjects).

For statistical analysis of AEs, the following analysis phases are defined for each subject.

Table 6.1: 1 Analysis phases for statistical analysis of AEs, and actual treatment for analysis of laboratory data, vital signs, ECG and local tolerability

| Study analysis phase | Label | Start | End |
|---|---|---|---|
| Screening <sup>1</sup> | Screening | Date of informed consent | Date/time of start of infusion |
| On treatment | Placebo,<br>1 mg BI,<br>10 mg BI,<br>25 mg BI,<br>50 mg BI,<br>100 mg BI or<br>200 mg BI<br>respectively | Date/time of start of infusion | 12:00 a.m. on day after last contact date |

<sup>&</sup>lt;sup>1</sup> See Section 6.7 for definition of baseline, which will be used in the statistical analyses of safety laboratory data, ECG and vital signs.

AE summary tables will present results for the on-treatment phase only. All AEs will be listed.

In AE tables in CTR Section 15.3 (but not in Appendix 16.1.13.1.8.1 and Appendix 16.1.13.1.8.2 AE tables), the following total will be provided in addition:

• "Total BI", defined as the total over all on-treatment phases involving BI

• "Total on-trt", defined as the total over all on-treatment phases, including placebo

Safety laboratory data, ECG, vital signs, PK, immunogenicity and exploratory biomarker parameters will be analysed based on treatment groups (Placebo, 1 mg BI, 10 mg BI, 25 mg BI, 50 mg BI, 100 mg BI or 200 mg BI) with clear differentiation between baseline (cf. Section 6.7) and on-treatment measurements. Measurements will be considered on-treatment, if they were taken within the on-treatment phases as defined in Table 6.1: 1.

More details on the technical implementation of these analyses are provided in the ADS Plan of this TSAP.

#### 6.2 IMPORTANT PROTOCOL DEVIATIONS

Consistency check listings (for identification of deviations from time windows) and a list of protocol deviations (e.g. deviations in drug administration, in blood sampling times, etc.) will be provided to be discussed at the Report Planning Meeting. At this meeting, it will be decided whether a discrepant data value can be used in analyses or whether it must be corrected in the clinical database. Each protocol deviation must be assessed to determine whether it is an important PD (IPD). For definition of IPDs, and for the process of identification of these, refer to the BI reference document "Identify and Manage Important Protocol Deviations (IPD)" (2) and the DV domain template.

If any IPDs are identified, they are to be summarised into categories and will be captured in the decision log. Categories which are considered to be IPDs in this trial are defined in the DV domain template. If the data show other IPDs, the definition in the DV domain template will be supplemented accordingly by the time of the Report Planning Meeting.

IPDs will be summarized and listed. Which kind of IPDs could potentially lead to exclusion from which analysis set is specified in the DV domain template. The decision on exclusion of subjects from analysis sets will be made at the latest at the Report Planning Meeting, after discussion of exceptional cases and implications for analyses.

Non-important COVID-19 related PDs will only be listed.

#### 6.3 SUBJECT SETS ANALYSED

The treated set (TS) and pharmacokinetic parameter analysis set (PKS) will be used as defined in the CTP, Section 7.3.

In addition, the following subject sets will be used:

All ECG analyses are performed on the TS, except for the exposure-response analyses, which are performed on the ECGPCS defined below.

• ECG PK concentration set (ECGPCS):

This subject set includes all subjects from the TS who provide at least one pair of a valid drug serum concentration and a corresponding (i.e. time-matched) ECG endpoint to be used in the exposure-response analyses. For placebo subjects, the

serum concentration is set to zero and hence always considered as valid. The decision whether a time deviation between PK blood sampling and ECG recording is acceptable (and thus whether the pair of values will be used) is to be made no later than at the RPM before data base lock. For subjects treated with active drug, the decision about concentration value validity needs to be made within the Clinical Pharmacology Group.



Table 6.3: 1 Subject sets analyzed

| | Subject sets | | |
|---|---|---|---|
| Class of endpoint | TS | PKS | ECGPCS |
| Primary endpoint | X | | |
| Secondary PK endpoints | | X | |
| Safety parameters | X | | |
| (except for exposure-response analyses of ECG data) | | | |
| Exposure-response analyses of<br>ECG data | | | X |
| | v | | |
| Demographic/baseline<br>characteristics | X | | |
| | X | | |

#### 6.5 POOLING OF CENTRES

This section is not applicable, because the study was performed in only one centre.

#### 6.6 HANDLING OF MISSING DATA AND OUTLIERS

CTP: "If a subject is removed or withdraws from the trial prior to the administration of trial medication, the data of this subject will not be entered in the case report form (CRF) and will not be reported in the clinical trial report (CTR). If a subject is removed or withdraws from the trial after the administration of trial medication, this will be documented and the reason for discontinuation must be recorded in the CRF. In addition, the data will be included in the CRF and will be reported in the CTR."

**CTP**: "It is not planned to impute missing values for safety parameters."

One exception where imputation might be necessary for safety evaluation is AE dates. Missing or incomplete AE dates are imputed according to BI standards (3).

If single cardiac cycles of an ECG are missing, the arithmetic mean for this single ECG will be computed with the reduced (1, 2 or 3) number of cardiac cycles. If replicate ECG recordings are missing, the arithmetic means per time point will be computed with the reduced number (1 or 2) of recordings.

For the classification of the on-treatment QTc/QT intervals into 'no new onset' / 'new onset' categories, the handling of missing value is described in <u>Additional Section 10.3.</u>

For the exposure-response analyses \_\_\_\_\_\_, missing serum concentration values with 'BLQ' in the comment field will be replaced by ½ LLOQ for subjects on active drug. For placebo subjects, the missing serum concentration values will be replaced by 0.

Missing data and outliers of PK data are handled according to BI standards ( $\underline{4}$ ) and ( $\underline{5}$ ).

**CTP**: "Pharmacokinetic parameters that cannot be reasonably calculated based on the available drug concentration-time data will not be imputed."

#### 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

In all analyses (except for analyses of ECG variables), baseline is defined as the last available value prior to start of infusion.

A centralised evaluation of 12-lead ECG recordings is performed at the time points specified in Table 6.7: 1

Table 6.7: 1 Time schedule of 12-lead ECG recordings with centralised evaluation

| Visit | Day | Planned time [hh:mm] - relative to start of infusion | Study phase |
|---|---|---|---|
| 2 | | -3:00 | Baseline |
| | | 00:30 | On-treatment |
| | | 01:00 | |
| | | 01:30 <sup>1</sup> | |
| | | 02:00 | |
| | | 03:00 | |
| | | 04:00 | |
| | | 06:00 | |
| | | 08:00 | |
| | 1 | 12:00 | |
| | 2 | 24:00 | |
| | | 34:00 | |
| | 3 | 48:00 | |

<sup>&</sup>lt;sup>1</sup> According to CTP flow chart, there is no time-matched PK sample for the ECG measurement at planned time 1:30. This ECG measurement will not be used in the exposure-response model, which will be applied to time matched pairs of ECG measurements and PK samples.

Three triplicate ECGs will be recorded as the baseline before drug administration, but only the first ECG of each of the 3 baseline triplicate will be transferred to the database. At all other time points, 1 triplicate ECG will be recorded, but only the first single ECG of the triplicate will be transferred to the database. The baseline value of an ECG variable is defined as the mean of the ECG variable values prior to drug administration.

Additional (unscheduled) ECGs may be recorded for safety reasons. These ECGs are assigned to the prior scheduled time point in the sponsor's database. Unscheduled ECGs (for safety reasons) will be transferred to the central ECG lab but will not be included into the statistical analysis of interval lengths.

For the exposure response analyses, pairs of ECG variables and corresponding serum concentrations will be built using the same planned time points, e.g., the HR change from baseline and the serum concentration measured at planned time 0:30 will build one pair. Whether a time deviation between PK blood sampling time and corresponding ECG recording is too big for a reliable assessment and the pair has to be excluded from the analysis will be decided no later than at the RPM.

Time windows are defined in Section 6.1 of the CTP. Adherence to time windows will be checked at the Report Planning Meeting.

#### 7. PLANNED ANALYSIS

The format of the listings and tables will follow the BI guideline "Reporting of clinical trials and project summaries" ( $\underline{6}$ ).

The individual values of all subjects will be listed. Listings will be sorted by treatment or sequence group, subject number and visit (if visit is applicable in the respective listing). AE listings will be sorted by assigned treatment (see Section 7.8.1 below for details). The listings will be contained in Appendix 16.2 (SDL) of the CTR.

The following standard descriptive statistical parameters will be displayed in summary tables of continuous variables:

N number of non-missing observations

Mean arithmetic mean SD standard deviation

Min minimum Median median Max maximum

For serum concentrations as well as for all PK parameters the following descriptive statistics will additionally be calculated:

CV arithmetic coefficient of variation

gMean geometric mean

gCV geometric coefficient of variation

For PK parameters the following descriptive statistics will additionally be calculated:

P10 10<sup>th</sup> percentile Q1 1<sup>st</sup> quartile Q3 3<sup>rd</sup> quartile P90 90<sup>th</sup> percentile

The data format for descriptive statistics of serum concentrations will be identical with the data format of the respective concentrations. The descriptive statistics of PK parameters will be calculated using the individual values with the number of decimal places as provided by the evaluation program. Then the individual values as well as the descriptive statistics will be reported with three significant digits in the CTR.

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category as well as the percentage (%) relative to the respective treatment group. Percentages will be rounded to one decimal place. The category missing will be displayed if and only if there actually are missing values. Percentages will be based on all subjects in the respective subject set whether they have non-missing values or not.

#### 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Only descriptive statistics are planned for this section of the CTR. These will be based on the TS.

#### 7.2 CONCOMITANT DISEASES AND MEDICATION

Concomitant diseases will be coded according to the most recent version of MedDRA. Concomitant medication will be coded according to the most recent version of the World Health Organisation – Drug Dictionary. Concomitant non-drug therapies will be coded according to the most recent version of MedDRA.

Only descriptive statistics are planned for this section of the CTR.

**CTP:** Previous and concomitant therapies will be presented per treatment group without consideration of time intervals and treatment periods.

A medication will be considered concomitant to a dose group, if it

- is ongoing at the time of study drug administration, or
- starts within the analysis phase of the respective treatment (see <u>Section 6.1</u> for a definition of treatments and analysis phases).

The relevance of the concomitant therapies to the evaluation of PK will be decided no later than at the RPM.

#### 7.3 TREATMENT COMPLIANCE

Treatment compliance will not be analyzed as a specific endpoint. Any deviations from complete intake will be addressed in the Report Planning Meeting (cf. Section 6.2) and described in the CTR.

#### 7.4 PRIMARY ENDPOINTS

#### 7.4.1 Primary analysis of the primary endpoints

Refer to <u>Section 7.8.1</u> for a description of the analysis of AEs, and in particular the analysis of the percentage of subjects with drug related AEs, which is the primary endpoint of this trial.

#### 7.5 SECONDARY ENDPOINTS

#### 7.5.1 Key secondary endpoints

This section is not applicable as no key secondary endpoint has been specified in the protocol.

#### 7.5.2 Secondary endpoints

The analysis of secondary endpoints will be based on the PKS.

#### 7.5.2.1 Secondary endpoint analysis

The PK endpoints will be assessed descriptively. The analysis of standard PK parameters is performed according to BI standards (4) [001-MCS-36-472 RD-01].

#### Exclusion of PK parameters

The ADS ADPP contains column variables APEXC and APEXCO indicating inclusion/exclusion (APEXC) of a PK parameter and an analysis flag comment (APEXCO). All analyses based on the PKS are based on PK parameter values which are not flagged for exclusion, i.e. with APEXC equal to "Included".

**CTP**: Serum concentration data and parameters of a subject which is flagged for exclusion will be reported with its individual values but will not be included in the statistical analyses.

#### Exclusion of PK concentrations

The ADS ADPC (PK concentrations per time-point or per time-interval) contains column variables ACEXC or ACEXCO indicating inclusion/exclusion (ACEXC) of a concentration and an analysis flag comment (ACEXCO). Exclusion of a concentration depends on the analysis flag comment ACEXCO. For example, if ACEXCO is set to "ALL CALC", the value will be excluded for all types of analyses based on concentrations. If ACEXCO is set to "DESC STATS" the value will be excluded from descriptive evaluations per planned time point/time interval. If ACEXCO contains the addition "TIME VIOLATION" or "TIME DEVIATION", the value can be used for further analyses based on actual times. If ACEXCO is set to "HALF LIFE", the value will be excluded from half-life calculation only; the value is included for all other analyses. Excluded concentration itself will be listed in the CTR associated with an appropriate flag.

Further details are given in "Noncompartmental Pharmacokinetic / Pharmacodynamic Analyses of Clinical Studies" (4) REF5 and "Description of Analytical Transfer Files and PK/PD Data Files" (5)



| 7.6.1 | Safety parameters |
|---|---|
| Safety end | dpoints and tolerability will be analysed as described in <u>Section 7.8</u> of this TSAP. |



#### 7.7 EXTENT OF EXPOSURE

Since only a single dose is administered per subject a listing will be sufficient to give account of the extent of exposure.

#### 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the TS, except for the exposure-response analysis which will be based on the ECGPCS.

#### 7.8.1 Adverse Events

AEs will be coded with the most recent version of MedDRA.

The analyses of AEs will be descriptive in nature. All analyses of AEs will be based on the number of subjects with AEs and not on the number of AEs.

For further details on summarization of AE data, please refer to "Analysis and Presentation of Adverse Event Data from Clinical Trials" (7) and "Handling of missing and incomplete AE dates" (3).

The analysis of AEs will be based on the concept of treatment emergent AEs. That means that all AEs will be assigned to screening or on-treatment phase as defined in <u>Section 6.1</u>. AEs will be analysed based on actual treatments, as defined in <u>Table 6.1: 1</u>.

An overall summary of AEs will be presented. This overall summary will comprise summary statistics for the class of AESIs.

**CTP:** Hepatic injury is considered an AESI in this trial. A hepatic injury is defined by the following alterations of hepatic laboratory parameters:

- An elevation of AST (aspartate transaminase) and/or ALT (alanine transaminase)  $\geq 3$  fold ULN combined with an elevation of total bilirubin  $\geq 2$  fold ULN measured in the same blood sample, or
- Aminotransferase (ALT, and/or AST) elevations  $\geq$ 10 fold ULN

The investigator had to classify on the eCRF whether an observed AE was an AESI or not.

According to ICH E3 (8), in addition to Deaths and Serious Adverse Events, 'other significant' AEs need to be listed in the clinical trial report. These will be any non-serious adverse event that led to an action taken with study drug (e.g. discontinuation or dose reduced or interrupted).

The frequency of subjects with AEs will be summarised by treatment, primary SOC and preferred term. AEs which were considered by the investigator to be drug related will be summarised separately. Separate tables will also be provided for subjects with SAEs and subjects with AESIs. AEs will also be summarized by maximum intensity.

The SOCs and preferred terms within SOCs will be sorted by descending frequency over all treatment groups.

For disclosure of AE data on ClinicalTrials.gov, the frequency of subjects with non-serious AEs occurring with an incidence of greater than 5 % (in preferred terms) will be summarised by treatment, primary SOC and preferred term. The frequency of subjects with SAEs will also be summarised.

For disclosure of AE data in the EudraCT register, the frequency of AEs, the frequency of non-serious AEs with an incidence of greater than 5 % (in preferred terms) and the frequency of SAEs will be summarized.

For support of lay summaries, the frequency of subjects with drug-related SAEs will be summarized by treatment, primary SOC and preferred term.

#### 7.8.2 Laboratory data

The analyses of laboratory data will be descriptive in nature and will be based on BI standards "Display and Analysis of Laboratory Data" (9).

Analyses will be based on normalised values, which means transforming to a standard unit and a standard reference range. The original values will be analysed if the transformation into standard unit is not possible for a parameter.

Descriptive statistics of laboratory values over time and for the difference from baseline (see <u>Section 6.7</u>) will be provided. Frequency tables of changes between baseline and last value on treatment with respect to the reference range will be presented.

Unscheduled measurements of laboratory data will be assumed to be repeat measurements of the most recent scheduled measurement (e.g. for follow-up or confirmation of a particular value). Therefore, unscheduled measurements will be assigned to the planned time point of the previous scheduled measurement. Descriptive statistics will be calculated by planned time point based on the worst value of the subject at that planned time point (or assigned to that planned time point).

Clinically significant abnormal laboratory values are only those identified either in the Investigator's comments or at the Report Planning Meeting at the latest. It is the Investigator's responsibility to decide whether a lab value is clinically significant abnormal or not.

Laboratory data will be compared to their reference ranges. Values outside the reference range as well as possibly clinically significant values will be highlighted in the listings. Possibly clinically significant laboratory values will be listed separately.

Clinically relevant findings in laboratory data will be reported as baseline conditions (prior to start of infusion) or as AEs (after start of infusion) if judged clinically relevant by the investigator, and will be analyzed as such.

#### 7.8.3 Vital signs

The analyses of vital signs (blood pressure and pulse rate) will be descriptive in nature. Descriptive statistics of vital signs over time and for the difference from baseline (see Section 6.7) will be provided.

Unscheduled measurements of vital signs will be assigned to planned time points in the same way as described above for laboratory data. However, for vital signs, descriptive statistics will be calculated by planned time point based on the last value of the subject at that planned time point (or assigned to that planned time point).

Clinically relevant findings in vital signs data will be reported as baseline conditions (prior to start of infusion) or as AEs (after start of infusion) if judged clinically relevant by the investigator, and will be analyzed as such.

#### 7.8.4 ECG

For continuous ECG and 12-lead ECG, abnormal findings, irrespective of whether they originate from central or local evaluation, will be reported as baseline conditions (prior to start of infusion) or as AEs (after start of infusion) if judged clinically relevant by the investigator.

Descriptive analysis of ECG endpoints will be based on the TS. The evaluation of the relationship between serum concentration and change in ECG endpoints (exposure-response analysis) will be based on the ECGPCS.

ECG measurements will not be included in the statistical analysis if one of the following applies:

- No date or time available for ECG measurement
- Pre-dose measurement done after start of infusion
- On-treatment measurement done before start of infusion
- Measurement is a repeated measurement

- More than 3 single ECGs (i.e., measurements from 4<sup>th</sup> single ECG onwards will not be included)
- Unscheduled measurements

#### Listing of individual data

For all quantitative endpoints, listings of individual data will be shown in Appendix 16.2. For QTcB and RR, only listings will be provided. Occurrences of notable findings will be flagged.

#### Categorical endpoints

For the categorical endpoints, frequency tables will be provided.

For all subjects with any notable finding in ECG intervals, a separate listing will be created as end-of-text display (based on the same display template as in Appendix 16.2), and the corresponding time profiles will be presented in figures.

#### Quantitative endpoints

Descriptive statistics (N, mean, SD, min, median, max) will be provided for the absolute values and changes from baseline over time of QTcF, HR, QT, PR and QRS. The time profiles of mean and SD for the changes from baseline on treatment will be displayed graphically by treatment.

#### Exposure-response analysis

For QTcF and HR changes from baseline, the relationship to the corresponding serum concentrations will be evaluated using a random coefficient model. For subjects in the ECGPCS, all time points with available ECG endpoints and valid time-matched drug serum concentrations will be included. For the handling of missing values, see <a href="Section 6.6">Section 6.6</a>.

The response variable will be the change from baseline in QTcF ( $\Delta$ QTcF). The placebo subjects will be included in the analysis, setting their serum concentrations to zero.

As a first step, it is investigated if there is a potential delayed or accelerated (e.g. due to metabolites) effect of the drug on QTcF. A general visual impression will be provided by overlaying time profiles of serum concentrations and QTcF changes from baseline (ΔQTcF). These figures will be generated for each subject (presented in the Statistical Appendix of the CTR), as well as for means per dose group (presented in the End-of-Text part of the CTR).

The relationship between BI 765080 serum concentrations and QTcF changes from baseline will be investigated in an exploratory manner using a random coefficient model to estimate the difference in mean QTcF change from baseline between BI 765080 and placebo and its 90% confidence interval at the geometric mean of  $C_{max}$  for each dose group. Additionally, the estimated overall slope with its 90% confidence interval will be provided. The used random coefficient model is based on a white paper from Garnett et. al. [R18-0143] (10) with  $\Delta$ QTcF as response variable, centered baseline QTcF and serum concentration as continuous

covariates, treatment, time and day as fixed categorical effects, and a random intercept and slope for each subject.

Restricted maximum likelihood estimation will be performed, and the Kenward-Roger method will be applied to adjust standard errors and estimate denominator degrees of freedom.

For more details refer to Section 10.4.

For visualization, a scatterplot of the BI 765080 serum concentration against the following individual QTcF values will be provided: For each subject on active treatment and each time point, subtract the mean value of all individual observed  $\Delta QTcF$  values from the placebo group for this time point from the individual observed  $\Delta QTcF$  value for this subject and time point. This results in estimates for "individual  $\Delta\Delta QTcF$ " values, which should only be used for plotting purposes. The corresponding regression line and its pointwise confidence bands as well as the geometric mean of  $C_{max}$  for each dose will additionally be displayed in the plot. The goodness of fit of the above model will be checked. The visual checks will include the inspection of concentration-QTcF quantile plots (see [R18-0143] (10)) and residual plots.

To check model assumptions, the conditional residuals will be plotted and presented in the Statistical Appendix of the CTR. In case of non-linearity or if there is evidence for a delayed effect, further models will be explored in order to better characterise the PK-ECG relationship (e.g. effect compartment models, non-linear models, etc.).

All of the above described graphical and statistical analyses for the exposure-reponse analysis will be also performed for HR in place of QTcF.

#### Appropriateness of heart rate correction methods of QT interval

To evaluate the appropriateness of the heart rate correction methods, the slope of the relationship of QTcF interval versus RR interval will be estimated separately for off-drug values and active treatment, by applying the random coefficient model described in Section 10.2 using the QTcF and RR variable values per time point. A scatterplot of QTcF vs RR including the overall regression lines will be included in the Statistical Appendix of the CTR. The resulting (fixed effect) slope together with two-sided 95% confidence intervals will be included in the footnote for this plot.

#### **7.8.5** Others

#### 7.8.5.1 Physical examination

Physical examination findings will be reported as relevant medical history/baseline condition (if a condition already exists before first administration of study treatment) or as AE (if condition emerges after first administration of study treatment) and will be summarized as such. No separate listing or analysis of physical examination findings will be prepared.

#### 7.8.5.2 Oral body temperature

Analysis of oral body temperature will be descriptive in nature.

## 7.8.5.3 Local tolerability assessment

Local tolerability (absence or presence of "swelling", "induration", "heat", "redness", "pain", or "other findings") will be summarized with counts and percentages overall (i.e. over all ontreatment time points, cf. Section 6.1) as well as by time point.

#### 7.8.5.4 Body weight

Body weight will only be listed.

# 8. TIMEPOINT OF RELEASE OF TREATMENT INFORMATION

The treatment information will be loaded into the trial database at trial initiation, i.e., the database will be handled open-label in accordance with the CTP.





Boehringer Ingelheim
TSAP for BI Trial No: 1450-0001
Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



Boehringer Ingelheim
TSAP for BI Trial No: 1450-0001
Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies





TSAP for BI Trial No: 1450-0001 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 11. **HISTORY TABLE**

History table Table 11: 1

| Version | Date<br>(DD-MMM-YY) | Author | Sections changed | Brief description of change |
|---|---|---|---|---|
| Final | 21-SEP-21 | | None | This is the final TSAP |